CLINICAL TRIAL: NCT04100148
Title: SyncAV Post-Market Trial
Acronym: SyncAV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10299
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Congestive Heart Failure
Keywords: SyncAV feature; CRT optimization; CRT non-responders; ECG optimization; Cardiac remodeling; CRT with SyncAV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SyncAV Arm (Experimental): Treatment Arm
  Interventions: Device: SyncAV programmed ON
- Fixed AV Delay Arm (Active Comparator): Control Arm
  Interventions: Device: Fixed AV delay

INTERVENTIONS:
Device: SyncAV programmed ON — For those subjects randomized to SyncAV programmed ON, sites will measure QRS duration with the subject's intrinsic rhythm (pacing OFF), at BiV pacing nominal settings, with various SyncAV programmed offsets, and at LV first 30 ms, RV first 30 ms and LV-only pacing with optimal SyncAV offsets. The site will then program the subject's device using the SyncAV offset that provided the narrowest QRS duration.
  Arms: SyncAV Arm
Device: Fixed AV delay — For those subjects randomized to the fixed AV delay arm, sites will measure QRS duration with the subject's intrinsic rhythm (pacing OFF) and at BiV pacing nominal settings. Sites will then program the subject's device using BiV pacing nominal settings.
  Arms: Fixed AV Delay Arm

SUMMARY:
The SyncAV Post-Market Trial is a prospective, randomized, multi-center trial performed to determine if cardiac resynchronization therapy (CRT) devices programmed with SyncAV ON improve long-term CRT response compared to devices programmed with conventional CRT through evaluation of changes in left ventricular (LV) reverse remodeling.

DETAILED DESCRIPTION:
The SyncAV Post-Market Trial is designed as a prospective, randomized, multi-center trial. The trial will require physicians to implant an Abbott CRT device and Abbott Quadripolar LV lead with any available right atrial and right ventricular leads. Sites will randomize subjects in a 1:1 ratio within 2 - 6 weeks post successful CRT implant: Arm 1 - SyncAV CRT programmed ON; Arm 2 - programmed fixed atrioventricular (AV) delay.

For those subjects randomized to SyncAV programmed ON, sites will measure QRS duration with the subject's intrinsic rhythm (pacing OFF), at biventricular (BiV) pacing nominal settings, with various SyncAV programmed offsets, and at LV first 30 ms, RV first 30 ms and LV-only pacing with optimal SyncAV offsets. The site will then program the subject's device using the SyncAV offset that provided the narrowest QRS duration.

For those subjects randomized to the fixed AV delay arm, sites will measure QRS duration with the subject's intrinsic rhythm (pacing OFF) and at BiV pacing nominal settings. Sites will then program the subject's device using BiV pacing nominal settings.

Sites will collect data at baseline (before CRT implant), randomization, and at 3-month, 6-month, and 12-month visits. For subjects randomized to the SyncAV ON arm, sites will optimize the SyncAV feature again at 3 months and 6 months in the same manner as the randomization visit.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to receive a new CRT implant or an upgrade (Abbott CRT device and Abbott Quadripolar LV lead) from an existing implantable cardioverter defibrillator/pacemaker implant with no more than 10% RV pacing at the last device interrogation, no prior LV lead placement, AND meet the following additional criteria:

   1. Mild to severe heart failure despite optimal medical therapy for at least 3 months prior to signing consent. Optimal medical therapy is defined as maximal tolerated dose of beta-blockers and a therapeutic dose of angiotensin-converting enzyme inhibitor, angiotensin receptor blocker, or aldosterone antagonist
   2. LVEF ≤ 35% based on a prior standard of care echocardiogram
   3. Left bundle branch block (LBBB) as documented on an ECG. Criteria for complete LBBB should include,

   i. QRS duration ≥ 120 ms ii. QS or rS pattern in leads V1 iii. mid-QRS notching or slurring in leads I, aVL, V5, and V6 iv. Absence of Q-wave in leads V5 and V6 d. Intact AV conduction (PR interval ≤ 280 ms on surface ECG)
2. At least 18 years old, or of legal age and willing and capable to give informed consent specific to each country and national laws
3. Willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

1. Recent myocardial infarction or unstable angina within 40 days prior to signing consent
2. Recent cardiac revascularization (angioplasty, stent or bypass graft) in the 4 weeks prior to signing consent or planned within 3 months following consent
3. Cerebrovascular accident or transient ischemic attack in the 3 months prior to signing consent
4. Any other therapeutic cardiovascular procedure (transcatheter aortic valve replacement, MitraClip, cardiac surgery, left atrial appendage closure, patent foramen ovale closure, or any ablation procedures) in the 3 months prior to signing consent
5. Permanent or persistent AF at the time of signing consent
6. Paroxysmal AF with at least one cardioversion within 60 days prior to signing consent
7. Prior CRT device implant
8. Prior His Bundle pacing implant or plan to have His Bundle pacing implant
9. Pregnant or breastfeeding at the time of signing consent
10. Incapacitated or unable to read or write
11. Undergone cardiac transplantation or have a classification of Status 1 for cardiac transplantation or consideration for transplantation during the study follow-up period
12. Life expectancy < 12 months due to any condition
13. Unavailable for at least 12 months of follow-up visits
14. Enrolled in or intend to participate in a clinical drug and/or device study during this clinical trial which could confound the results of this trial as determined by Abbott

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1686 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in left ventricular end systolic volume (LVESV) between baseline and 12 months | 12 months following trial randomization
  Reduction of LVESV as a continuous variable from baseline to 12 months compared between subjects in the SyncAV and fixed AV delay arms.

SECONDARY OUTCOMES:
Percentage of CRT Responders at 12 months | 12 months following trial randomization
  Percentage of subjects classified as CRT responders after 12 months of follow-up compared between subjects in the SyncAV and fixed AV delay arms, as measured by LVESV reduction of at least 15% compared to baseline.
Reduction in LVESV in female subjects between baseline and 12 months | 12 months following trial randomization
  Reduction of LVESV as a continuous variable from baseline to 12 months compared between female subjects in the SyncAV and fixed AV delay arms.
Percentage of female subjects classified as CRT Responders at 12 months | 12 months following trial randomization
  Percentage of female subjects classified as CRT responders after 12 months of follow-up compared between female subjects in the SyncAV and fixed AV delay arms, as measured by LVESV reduction of at least 15% compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Varma, MD, Principal Investigator — The Cleveland Clinic
Locations (104):
- United States (30):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - Comprehensive Cardiovascular, Bakersfield, California
  - Cardiovascular Consultants Heart Center, Fresno, California
  - USC University Hospital, Los Angeles, California
  - Colorado Heart & Vascular, P.C., Lakewood, Colorado
  - Shands at the University of Florida, Gainesville, Florida
  - Heart Rhythm Solutions, Hollywood, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CHI St. Luke's Health Baylor College of Medicine Med. Ctr., Houston, Texas
  - Memorial Katy Cardiology Associates, Houston, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Heart Rhythm Associates, Shenandoah, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Universitätsklinik Graz, Graz, Styria, Austria
- Hopital Erasme, Brussels, Belgium
- Canada (16):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Hopital du Sacre-Coeur de Montreal, Montreal, Montreal
  - HSC, Eastern Health, St. John's, Newfoundland and Labrador
  - QE II Health Sciences, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - Cardiac Arrhythmia Research Group Inc. (CARGI), Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - McGill University Health Centre General Hospital, Montreal, Quebec
  - CHUS Fleurimont, Sherbrooke, Quebec
  - Royal Alexandra Hospital, Edmonton
  - CHUM, Montreal
  - Institut de Cardiologie de Quebec (Hôpital Laval), Québec
- China (3):
  - Tianjin Chest Hospital, Tianjin, Heping
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
- Helsinki University Central Hospital (HYKS), Helsinki, Finland
- France (5):
  - CHU Rangueil Toulouse, Toulouse, Midi-Pyrenees
  - CHRU Hopital de Pontchaillou, Rennes
  - St-Etienne CHU, Saint-Priest-en-Jarez
  - Hopital Henri Mondor, Créteil, Île-de-France Region
  - CHR de La Reunion - Site du CHFG, Saint-Denis, Île-de-France Region
- Germany (3):
  - Klinikum der Ruprecht-Karls-Universität Heidelberg, Heidelberg, Bad-wur
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden, Saxony
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
- The University of Hong Kong (Queen Mary Hospital), Hong Kong, Hong Kong
- India (6):
  - Asian Institute of Gastroenterology (AIG) Hospital, Hyderabad, Andprad
  - Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Apollo Hospitals, Bangalore, Bangalore, Karnataka
  - Narayana Institute of Cardiac Sciences, Bommasandra, Bangalore, Karnataka
  - Medanta - The Medicity Hospital, Gūrgaon
  - Max Super Specialty Hospital, New Delhi
- Italy (4):
  - Mater Dei Hospital, Bari, Apulia
  - Azienda Ospedaliera Di Venere, Carbonara, Apulia
  - Azienda Ospedaliera Universitaria MaterDomini, Catanzaro, Calabria
  - Azienda Ospedaliera S. G. Moscati, Avellino
- Japan (4):
  - Chiba University, Chiba, Chiba
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagwa
- Amsterdam Academic Medical Centre (AMC), Amsterdam, Noord-h, Netherlands
- Poland (2):
  - Scanmed SA, Krakow, Lesrpld
  - Szpital Kliniczny Przemienienia Panskiego UM w Poznaniu, Poznan
- Santa Maria Hospital, Lisbon, Portugal
- Arrhythmia Group LLC, Ponce, Puerto Rico
- Meshalkin National Medical Research Center, Novosibirsk, Siberia, Russia
- Saudi Arabia (3):
  - King Fahad Armed Forces Hospital, Jeddah, Mecca Region
  - King Faisal Specialist Hospital (KFSH), Riyadh, Riyadh Region
  - King Fahad Medical City, Riyadh
- Clinical Center of Serbia - Pacemaker Center, Belgrade, Serbia
- South Korea (7):
  - Sejong Hospital, Bucheon-si, Sudogwn
  - Keimyung University Dongsan Medical Center, Daegu, Sudogwn
  - Seoul National University Bundang Hospital, Seongnam, Sudogwn
  - Samsung Medical Center, Seoul, Sudogwon
  - Keimyung University Dongsan Medical Center, Daegu
  - Asan Medical Centre, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (6):
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Clínic de Barcelona, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - Hospital Puerta de Hierro - Hospital Universitario, Madrid
  - HCU Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
- Karolinska University Hospital, Solna, Stockholm, Sweden
- Taichung Veterans General Hospital, Taichung, Taiwan
- Phramongkutklao Hospital, Bangkok, Central Thailand, Thailand
- United Kingdom (3):
  - Southampton University Hospital, Southampton, Soeast
  - John Radcliffe Hospital, Oxford, South East England
  - The Royal Sussex County Hospital, Brighton

IPD SHARING:
Plan to Share IPD: No